CLINICAL TRIAL: NCT00917423
Title: Physical Activity in Anorexia Nervosa: Characteristics and Clinical Significance
Brief Title: Characteristics and Importance of Physical Activity in Women With Anorexia Nervosa
Status: Completed | Type: Observational
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: #5544/#6624R; R01MH083795 (NIH); DATR A2-AIM (Other Grant/Funding Number: DATR A2-AIM)
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-05

CONDITIONS: Eating Disorders
Keywords: Anorexia Nervosa; Exercise; Physical Activity
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Inpatients with anorexia nervosa: Hospital inpatients with anorexia nervosa
- Normal weight controls: Healthy, normal-weight volunteers

SUMMARY:
This study will determine the importance and the level of physical activity among women with anorexia nervosa, both during inpatient treatment and 1 year after hospital discharge.

DETAILED DESCRIPTION:
Anorexia nervosa is a disorder that causes people to maintain an unhealthily low body weight, often through eating too little or exercising too much. Treatment for anorexia nervosa often begins with a supervised program for raising a person's weight to a healthy level. This study will monitor activity levels during inpatient treatment and for 1 year after hospital discharge in order to determine the impact of physical activity on weight gain during anorexia treatment.

Participation in this study will last until 1 year after participants are discharged from inpatient treatment for anorexia nervosa. Discharge is based on each person's progression in treatment and may vary among participants. During the study, participants will have their activity monitored two or three times-at low weight, at 90% of ideal body weight (IBW), and, if the participant is living near the study clinic, within 6 weeks after discharge from the hospital. Two monitoring devices will be attached to participants continuously for 48 hours for the first two assessments and for 72 hours for the third. The first device is a SenseWear armband, which is a wireless monitor strapped to the back of the upper arm that measures body movement and body temperature. The second is an Intelligent Device for Energy Expenditure and Activity (IDEEA) monitor, which consists of five sensors that will be taped to each participant's feet, thighs, and chest. The device measures activity levels and energy expenditure. Participants will complete a blood draw within 1 week of completing activity monitoring assessments. Participants will also complete a computer "work" task at two time points-at 75% of IBW and at 90% of IBW. This task will last 40 minutes and will involve tapping a keyboard in order to earn rewards. Adult participants will also complete a dual X-ray absorptiometry (DXA) test to assess body composition when 90% IBW is reached.

Follow-up assessments will occur 1, 2, 4, and 8 months after discharge. These will involve a phone call or in-person visit in which health, body weight, and eating disorder symptoms are discussed. One year after discharge, participants will attend an in-person assessment that will involve completing questionnaires and an interview. Healthy participants will be recruited as a control group, and these participants will complete one session of activity monitoring, one blood draw, and self-rating forms without follow-up measurements.

ELIGIBILITY:
Inclusion Criteria:

* Anorexia nervosa (except amenorrhea), as defined by DSM-IV
* Medically and psychiatrically stable

Exclusion Criteria:

* Significant current or past medical illness, including diabetes mellitus and heart disease
* Current or lifetime history of schizophrenia, bipolar disorder, or other psychotic disorder, as defined by DSM-IV-TR
* Suicidal ideation or suicidal behavior within the past 3 months
* Drug or alcohol abuse in last 6 months
* Taking psychotropic medication
* Pregnant

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients with anorexia nervosa participating in an inpatient treatment program
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2009-02; Primary Completion 2015-02 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in weight | Measured at baseline and 1 year after hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: B. Timothy Walsh, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- See also: Click here for more information on the Columbia Center for Eating Disorders — http://www.columbiacenterforeatingdisorders.org